CLINICAL TRIAL: NCT05445362
Title: Evaluation of the Efficacy of Diode Laser in Maturogenesis of Immature Teeth With Necrotic Pulps: A Preliminary Randomized Controlled Trial
Brief Title: Efficacy of Diode Laser in Maturogenesis of Immature Teeth With Necrotic Pulps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Hassan (Other)
Responsible Party: Sponsor-Investigator, Reham Hassan, Assoc. Prof. Dr Reham Hassan, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 145
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Effects of the Elements
Keywords: Diode Laser, Revascularization, Immature Necrotic Teeth.

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Thirteen teeth were disinfected by triple antibiotic paste then revascularization was done using the standard method.
  Interventions: Drug: Triple antibiotic paste disinfection; Procedure: revascularization using the standard method "Blood Clot"
- Group II (Active Comparator): Thirteen teeth were Laser disinfected; revascularization was done using the standard method.
  Interventions: Device: Diode laser disinfection; Procedure: revascularization using the standard method "Blood Clot"
- Group III (Active Comparator): Thirteen teeth were disinfected by triple antibiotic paste then revascularization was done using the standard method followed by diode laser bio-stimulation.
  Interventions: Device: Diode Laser bio-stimulation.; Drug: Triple antibiotic paste disinfection; Procedure: revascularization using the standard method "Blood Clot"

INTERVENTIONS:
Device: Diode laser disinfection — - Disinfection with parameter of Power: 1.5 watt, Mode: pulse: SP: Ton=10ms; Toff10ms 50Hz (50% pulse mode), for 5 seconds in spiral movement in apical to coronal direction no stop with non-initiated endodontic tip 200 micron diameter and 15 mm length three times. Irrigation with NaOCl, irradiation with the laser, then irrigation with E.D.T.A and irradiation with the laser, for three times then final rinse with distilled water with paper point dryness in between irrigations.
  Arms: Group II
Device: Diode Laser bio-stimulation. — - The diode laser bio-stimulation with Wiser Diode Laser, Irradiation of the periapical area from the labial mucosal surface, day after day "day on-day off" for one week, two sessions will be applied at the same day with two hours interval, first session immediately after filing (blood induction), with flat top hand piece , diameter 1cm at a distance between 0 and 105 cm, at 1 watt power for 50s with CW "continues mode" in order to obtain the 5 J/cm2 fluence.
  Arms: Group III
Drug: Triple antibiotic paste disinfection — -The root canals will be copiously and slowly irrigated with 20 ml of 1.5% (17) sodium hypochlorite (NaOCl) solution for 5 minutes alternatively with 20 ml of 17% ethylene diamine tetra acetic acid (E.D.T.A) solution for 5 minutes with intermediated rinse of distilled water with paper point dryness in between irrigations. The triple antibiotic paste will be prepared using metronidazole , ciprofloxacin and doxycycline . The doxycycline capsule content will be evacuated in a sterile mortar; a tablet of metronidazole and a tablet of ciprofloxacin will be crushed and ground into homogenous powder in the same mortar using a pestle. Saline drops will be added and mixed using the pestle until a creamy paste achieved . The canals Will be dried with paper points and medicated with triple antibiotic paste; the access cavity will be sealed with intermediate restorative material (I.R.M) .
  Arms: Group I; Group III
Procedure: revascularization using the standard method "Blood Clot" — - The root canal Will be over-instrumented using finger plugger size #25 to encourage bleeding up to cemento-enamel junction. The sterile finger plugger size # 25 will be used with sharp strokes into the periapical tissue beyond the apex until bleeding becomes evident at the cervical portion of the canal. Blood column will be left 10 minutes to clot covered by sterile cotton, a collagen orifice plug "Collagen plugs" will be used as matrix against mineral trioxide aggregate (M.T.A) condensation, M.T.A will be mixed according to the manufacturer's instructions and carried to the cavity with M.T.A carrier (Dovgan M.T.A Carrier) , and then compacted using wet cotton roll on pluggers (S- Kondenser) . Finally the cavity will be restored with a glass ionomer base and light cure composite resin .
  Other Names: Blood Clot revascularization method

SUMMARY:
Recruited patients with immature permanent maxillary anterior teeth with non-vital pulp, and periapical radiolucency, age ranging from 8 to16 years old were randomly allocated into three groups (n=13): Group I, disinfected using the triple antibiotic paste, Group II, disinfection was done using diode laser, and Group III, were disinfected using the triple antibiotic paste, diode laser was used for biostimulation. All groups were evaluated for the increase in root length and thickness and decrease in apical diameter at baseline, 3, 6, 9, and 12 months after treatment

DETAILED DESCRIPTION:
* The investigator recruited patients who are found eligible to the criteria then randomly allocated into three groups (n=13)
* Group I: thirteen teeth were disinfected by triple antibiotic paste then revascularization was done using the blood clot method.
* Group II: thirteen teeth were Laser disinfected; revascularization was done using the the blood clot method.
* Group III: thirteen teeth were disinfected by triple antibiotic paste then revascularization was done using the the blood clot method followed by diode laser bio-stimulation.
* periapical x rays was taken at baseline, 3, 6, 9, and 12 months after treatment for the increase in root length and thickness, decrease in apical diameter evaluation

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Immature permanent maxillary anterior teeth.
* Non vital pulp.
* patents age between 8-16 years.
* Both sexes.
* Restorable teeth.
* No internal or external root resorption.
* No horizontal or vertical root fracture
* Radiographic periapical radiolucency
* No history of previous endodontic treatment of the tooth.

Exclusion Criteria:

* Medically compromised patients
* Previous endodontic therapy of the affected tooth.
* Teeth diagnosed with vital pulp.
* Teeth with periodontal pocket more than 3mm deep.
* Teeth with caries below the bony level (non-restorable tooth).
* Mature teeth with complete apices.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
The change in root length evaluation | at baseline, 3, 6, 9, and 12 months after treatment
  Numerical using Image-J analysis software for radiographs standardization and measuring in mm, the percentage of change in length will be calculated by subtracting the 12 m length from the baseline , 3, 6, 9 months lengths divided by the baseline, 3, 6, 9 months length multiplying the value by 100
  - post length - pre length / pre length x 100

SECONDARY OUTCOMES:
The change in root thickness | At base line , 3, 6, 9, and 12 month after treatment
  Measurements in mmm using Image-J analysis software for radiographs standardization and measuring, the percentage of change in root width will be calculated by subtracting the 12 m length from the baseline , 3, 6, 9 months lengths divided by the baseline, 3, 6, 9 months widths multiplying the value by 100
The change in apical diameter | At base line, 3, 6, 9, and 12 month after treatment
  Measurements in mmm using Image-J analysis software for radiographs standardization and measuring, the percentage of apical diameter size change will be calculated as follows
  - pre diameter - post diameter / pre diameter X 100 , to get the percentage of apical diameter change with the deferent time changes "baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Reham Hassan, Assoc, prof, Study Director — Minia University
Locations (1):
- Faculty of Oral and dental medicine, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF